CLINICAL TRIAL: NCT02774707
Title: Comparing the Quality of Topical Autologous Serum in Different Etiologies of Dry Eye Syndrome
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201511091RINB
Record Dates: First submitted 2016-01-10; First posted 2016-05-17 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-12

CONDITIONS: Dry Eye Syndrome
Keywords: Dry eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Human autologous serum is commonly used in the treatment of dry eye disease. However, different patients may have different effect with autologous serum treatment. We would like to find if different autologous serum had different component of cytokines in different etiologies of dry eye.

DETAILED DESCRIPTION:
Dry eye is an important issue in the filed of ophthalmology and has great influence on the quality of life in many patients. Traditional treatment was mainly focused on artificial tear supplement. Inflammatory factors are identified in the recent days and are thought to play an important role in the etiology of dry eye. Anti-inflammatory agent like topical immunosuppressant has become another choice in the treatment of dry eye.

Conventional artificial tear has similar biochemical features and osmolarity with natural tear but lacks the anti-inflammatory cytokines. Therefore, autologous serum has been applied as a substitute of natural tear because it has more anti-inflammatory cytokines. Clinical trials have shown that autologous serum drops improve ocular irritation symptoms, and conjunctival and corneal dye staining in dry eye.

However, in the manufacture of autologous serum, it is hard to standardize every step and control quality. What's more, the patient may have different etiology of dry eye, including primary Sjogren's syndrome, secondary Sjogren's syndrome, other autoimmune disease, or ocular graft versus host disease. The etiology of dry eye may have different response to autologous serum. However, we don't know if the autologous serum from different patients' have different components and the different components of cytokines may have different treatment efficacy. This is what we want to know in this study.

Since human autologous serum is needed for cytokine analysis, we proposed this project to collect human serum from volunteers。

ELIGIBILITY:
Inclusion criteria

* Healthy volunteer control without ophthalmic history
* Patients with Primary Sjogren's syndrome: according to the classification of American European Consensus Group of rheumatologist and Ophthalmologists,
* Patient with Secondary Sjogren's syndrome: Sjogren's syndrome associated with systemic lupus erythematosus, systemic sclerosis (scleroderma), rheumatoid arthritis, mixed connective tissue disease, inflammatory muscle disease, autoimmune liver disease, and autoimmune thyroid disease
* Ocular graft versus host disease
* Volunteers with dry eye symptoms but not diagnosed with primary Sjogren's syndrome, secondary Sjogren's syndrome and ocular graft versus host disease

Exclusion criteria

* Patients who decline to receive the venipuncture for blood sampling.
* Patients younger than 20 years old or older than 80 years old.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Patients who need autologous human serum as treatment of dry eye disease
  2. Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Epidermal growth factor concentration in human autologous serum from different etiologies of dry eye | 1 year
  We would measure Epidermal growth factor concentration (ng/ml) by ELISA according to the manufactures instruction.
  We plan to collect 40 patients from different groups.
Transforming growth factor beta (ng/ml) concentration in human autologous serum from different etiologies of dry eye | 1 year
  We would measure Transforming growth factor beta (ng/ml) by ELISA according to the manufactures instruction.
  We plan to collect 40 patients from different groups.
Fibronectin (ug/ml) concentration in human autologous serum from different etiologies of dry eye | 1 year
  We would measureFibronectin (ug/ml) concentration by ELISA according to the manufactures instruction.
  We plan to collect 40 patients from different groups.
Hyaluronic acid (ug/ml) concentration in human autologous serum from different etiologies of dry eye | 1 year
  We would measure Hyaluronic acid (ug/ml) concentration by ELISA according to the manufactures instruction.
  We plan to collect 40 patients from different groups.

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Li Chen, Principal Investigator — ational Taiwan University Hospital, Ophthalmology Department
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided